CLINICAL TRIAL: NCT04553354
Title: Evaluation of Safety and Efficacy of Cortical Resections for Seizure Control for Patients With Drug Resistant Epilepsy
Brief Title: Cortical Resections in Drug Resistant Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Ammar, principal investigator, Assiut University
Other Study IDs: epilepsy surgery
Record Dates: First submitted 2020-09-09; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Epilepsy Surgery; Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cortical resections — is the removal of the epileptic focus either temporal or extra temporal area

SUMMARY:
The aim of the study is to evaluate safety and efficacy of epilepsy surgery in the form of cortical resections in patients with refractory epilepsy and to review outcomes of resection procedures in focal epilepsy.

DETAILED DESCRIPTION:
Nearly one-third of epilepsy patients are refractory/resistant to medical treatment . Refractory or drug-resistant epilepsy is defined as resistance to treatment with two appropriately chosen and tolerated antiepileptic drugs (AED) . Nevertheless, epilepsy surgery is an effective alternative treatment for some patients as it suggests seizure freedom . During the past 3 decades, surgery has found more acceptance as an option for drug-resistant epilepsy . Developments made in surgical techniques (cortical resections) have significantly increased the effectiveness and safety of these techniques; as such techniques have been demonstrated to improve seizure control/freedom outcomes and enhanced quality of life in patients . Neuro imaging developments with the introduction of positron emission tomography (PET), magnetic resonance imaging (MRI), functional MRI, single-photon emission computed tomography (SPECT), and magneto encephalography, electroencephalography and neuronavigation have facilitated the presurgical evaluation of patients, thus providing the lesion-directed surgeries more possible , also reducing the number and severity of complications . Complications of epilepsy surgery including failure to stop seizures and neuropsychological, psychosocial, or psychiatric impairment are still difficult to define, and there is no universal consensus in this regard .

This technique characterized by :

• Once the epilepsy focus is located by using interpretation and collection of data from functional MRI, EEG long term video and clinical findings, the specific surgery involved in treatment is decided on. The type of surgery depends on the location of the seizure focal point. Surgeries for epilepsy treatment include, but are not limited to, the following types: temporal lobe resection, ground temporal and extra temporal resection, parietal resection, occipital resection, frontal resection, extra temporal resection.

ELIGIBILITY:
Inclusion Criteria:

* All patients with focal epilepsy who are refractory to medical treatment.
* Patients accept surgical maneuver

Exclusion Criteria:

* Epileptic patients responding to medical treatment.
* Patients refusing surgical intervention.
* Patients unfit for brain surgery.
* Multi focal or generalized seizures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with focal epilepsy not responding to medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-09-10 (Estimated); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-11-10 (Estimated)

PRIMARY OUTCOMES:
control of focal epilepsy in drug resistant epileptic patients | baseline
  seizure freedom after cortical resections will be measured by angel classification
decrease incidence of drug adverse effects in drug resistant focal epilepsy | baseline
  the well known adverse effects of AEDs that are mentioned in literature as affection of the liver and kidney will be measured preoperatively by kidney function and liver function tests to detect if it is normal or not

SECONDARY OUTCOMES:
change quality of life of patients with drug resistant epilepsy | baseline
  changing quality of life of those patients as regards socioeconomic status of the patients if they get a jop or not and remain in his jop or not and the financial status improved or not and all of this will be mentioned by the patients in follow up in out patient clinic

REFERENCES:
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Background] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Background] Engel J Jr, McDermott MP, Wiebe S, Langfitt JT, Stern JM, Dewar S, Sperling MR, Gardiner I, Erba G, Fried I, Jacobs M, Vinters HV, Mintzer S, Kieburtz K; Early Randomized Surgical Epilepsy Trial (ERSET) Study Group. Early surgical therapy for drug-resistant temporal lobe epilepsy: a randomized trial. JAMA. 2012 Mar 7;307(9):922-30. doi: 10.1001/jama.2012.220. PMID 22396514
- [Background] Engel J Jr, Wiebe S, French J, Sperling M, Williamson P, Spencer D, Gumnit R, Zahn C, Westbrook E, Enos B; Quality Standards Subcommittee of the American Academy of Neurology; American Epilepsy Society; American Association of Neurological Surgeons. Practice parameter: temporal lobe and localized neocortical resections for epilepsy: report of the Quality Standards Subcommittee of the American Academy of Neurology, in association with the American Epilepsy Society and the American Association of Neurological Surgeons. Neurology. 2003 Feb 25;60(4):538-47. doi: 10.1212/01.wnl.0000055086.35806.2d. PMID 12601090
- [Background] Cukiert A, Rydenhag B, Harkness W, Cross JH, Gaillard WD; Task Force for Pediatric Epilepsy Surgery for the ILAE Commissions of Pediatrics and Surgical Therapies. Technical aspects of pediatric epilepsy surgery: Report of a multicenter, multinational web-based survey by the ILAE Task Force on Pediatric Epilepsy Surgery. Epilepsia. 2016 Feb;57(2):194-200. doi: 10.1111/epi.13292. Epub 2016 Jan 8. PMID 26749250
- [Background] Berg AT. Epilepsy: Efficacy of epilepsy surgery: what are the questions today? Nat Rev Neurol. 2011 Jun 8;7(6):311-2. doi: 10.1038/nrneurol.2011.73. PMID 21654716
- [Background] Tellez-Zenteno JF, Dhar R, Wiebe S. Long-term seizure outcomes following epilepsy surgery: a systematic review and meta-analysis. Brain. 2005 May;128(Pt 5):1188-98. doi: 10.1093/brain/awh449. Epub 2005 Mar 9. PMID 15758038
- [Background] Malmgren K, Sullivan M, Ekstedt G, Kullberg G, Kumlien E. Health-related quality of life after epilepsy surgery: a Swedish multicenter study. Epilepsia. 1997 Jul;38(7):830-8. doi: 10.1111/j.1528-1157.1997.tb01471.x. PMID 9579911
- [Background] Engel J Jr. Why is there still doubt to cut it out? Epilepsy Curr. 2013 Sep;13(5):198-204. doi: 10.5698/1535-7597-13.5.198. PMID 24348103
- [Background] A global survey on epilepsy surgery, 1980-1990: a report by the Commission on Neurosurgery of Epilepsy, the International League Against Epilepsy. Epilepsia. 1997 Feb;38(2):249-55. doi: 10.1111/j.1528-1157.1997.tb01105.x. No abstract available. PMID 9048680
- [Background] Rafael H. Surgical and neurological complications in a series of 708 epilepsy surgical procedures. Neurosurgery. 1998 Mar;42(3):675-6. doi: 10.1097/00006123-199803000-00048. No abstract available. PMID 9527007
- [Background] Cascino GD, Sharbrough FW, Trenerry MR, Marsh WR, Kelly PJ, So E. Extratemporal cortical resections and lesionectomies for partial epilepsy: complications of surgical treatment. Epilepsia. 1994 Sep-Oct;35(5):1085-90. doi: 10.1111/j.1528-1157.1994.tb02559.x. PMID 7925156
- [Background] Vakharia VN, Duncan JS, Witt JA, Elger CE, Staba R, Engel J Jr. Getting the best outcomes from epilepsy surgery. Ann Neurol. 2018 Apr;83(4):676-690. doi: 10.1002/ana.25205. Epub 2018 Apr 10. PMID 29534299